CLINICAL TRIAL: NCT03101618
Title: The Prevalence of Animal Allergy and Sensitization to Animal Allergen Among Participants in International Symposium of Korean Association for Laboratory Science and Companion Animal Exhibition
Brief Title: Animal Allergy in Korean Pet Owners, Pet-related Industry Workers, and Laboratory Animal Reseachers
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin Lee, MD, Assistant professor, Gachon University Gil Medical Center
Other Study IDs: GBIRB2016-155
Record Dates: First submitted 2017-03-29; First posted 2017-04-05 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis; Urticaria; Asthma
Keywords: allergen; allergy; pet
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic; Urticaria; Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Allergic LAR: Laboratory animal researchers who experienced allergic symptom during exposure to laboratory or pet animals
  Interventions: Other: Animal allergy
- Non-allergic LAR: Laboratory animal researchers who did not experience allergic symptom during exposure to laboratory or pet animals
  Interventions: Other: Non-animal allergy
- Allergic PO: Pet owners who experienced allergic symptom during exposure to pet animals
  Interventions: Other: Animal allergy
- Non-allergic PO: Pet owners who did not experience allergic symptom during exposure to pet animals
  Interventions: Other: Non-animal allergy
- Allergic PIW: Allergic pet-related industry workers who experienced allergic symptom during exposure to pet animals
  Interventions: Other: Animal allergy
- Non-allergic PIW: Allergic pet-related industry workers who did not experience allergic symptom during exposure to pet animals
  Interventions: Other: Non-animal allergy

INTERVENTIONS:
Other: Animal allergy — Allergic symptom occurs during exposure to laboratory or pet animal
  Groups: Allergic LAR; Allergic PIW; Allergic PO
Other: Non-animal allergy — Allergic symptom does not occur during exposure to laboratory or pet animal
  Groups: Non-allergic LAR; Non-allergic PIW; Non-allergic PO

SUMMARY:
The investigators surveyed the prevalence of animal allergy and sensitization to animal allergen among participants in international symposium of Korean association for laboratory science (laboratory animal researchers) and companion animal exhibition (pet owner and pet-related industry workers).

DETAILED DESCRIPTION:
The investigators enrolled participants in international symposium of Korean association for laboratory science (laboratory animal researchers) and pet animal exhibition (pet owner and pet-related industry workers) after informed consents. Subjects were asked to response to questionnaires regarding their age, gender, comorbid allergic disease, family history of allergy, pet or laboratory animal, exposure time, allergic symptoms during exposure to animals. Subjects underwent skin prick test with animal allergens and other inhalant allergens.

ELIGIBILITY:
Inclusion Criteria:

* Participants in international symposium of Korean association for laboratory science and companion animal exhibition from whom informed consents were obtained.

Exclusion Criteria:

* Subjects who reject enrollment into this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in international symposium of Korean association for laboratory science and companion animal exhibition
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2016-11-27 (Actual); Study Completion 2016-11-27 (Actual)

PRIMARY OUTCOMES:
Skin reactivity to animal allergens | The day of survey
  Positivity to animal allergens in skin prick test

SECONDARY OUTCOMES:
Skin reactivity to other inhalant allergens | The day of survey
  Positivity to other inhalant allergens in skin prick test
The prevalance of cormobid allergy | The day of survey
  The prevalance of allergic rhinitis, allergic conjunctivitis, asthma, urticaria, atopic dermatitis, contact dermatitis, food allergy, drug allergy
Duration of animal exposure | The day of survey
  Duration of laboratory or pet animal exposure (months)
Animal contact time | The day of survey
  Animal contact time including direct contact and spatial sharing (min/day)
Residence of animal | The day of survey
  Residence of animal (cage, bedroom, not bedroom but at home, outside)
Site of animal defecation | The day of survey
  Site of animal defecation (outside, predetermined place at home, anywhere at home)
Laboratory or pet animal | The day of survey
  Laboratory or pet animal which subject contacts
Severity of allergic symptom | The day of survey
  Severity of allergic symptom (using visual analog scale) during exposure to animal
Duration of allergic symptom | The day of survey
  Duration of allergic symptom during exposure to animal (min)
Frequency of house cleaning, bed cleansing, animal haircut, and animal hair removal from their garmet | The day of survey
  Frequency of house cleaning, bed cleansing, animal haircut, and animal hair removal from their garmet in pet owners and pet-related industry workers
Use of medical service | The day of survey
  Use of medical service including prescription and immunotherapy for animal allergy
Perception of animal allergy, its avoidance and immunotherapy | The day of survey
  Agreement score (visual analog scale) to "Allergic symptom occurs during exposure to animal", "Avoidance can reduce or prevent from allergic symptom", "Immunotherapy can mitigate allergic symptom during exposure to animal"

CONTACTS AND LOCATIONS:
Overall Officials: Sang Pyo Lee, MD, Study Chair — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park YB, Mo EK, Lee JY, Kim JH, Kim CH, Hyun IG, Choi JH. Association between pet ownership and the sensitization to pet allergens in adults with various allergic diseases. Allergy Asthma Immunol Res. 2013 Sep;5(5):295-300. doi: 10.4168/aair.2013.5.5.295. Epub 2013 Jun 25. PMID 24003386
- [Result] Moghtaderi M, Farjadian S, Abbaszadeh Hasiri M. Animal allergen sensitization in veterinarians and laboratory animal workers. Occup Med (Lond). 2014 Oct;64(7):516-20. doi: 10.1093/occmed/kqu097. Epub 2014 Aug 7. PMID 25104279
- [Result] Krakowiak A, Wiszniewska M, Krawczyk P, Szulc B, Wittczak T, Walusiak J, Palczynski C. Risk factors associated with airway allergic diseases from exposure to laboratory animal allergens among veterinarians. Int Arch Occup Environ Health. 2007 May;80(6):465-75. doi: 10.1007/s00420-006-0153-0. Epub 2006 Oct 5. PMID 17021840